CLINICAL TRIAL: NCT01323699
Title: Increasing Access and Implementation of Behavioral Treatments for Anxiety and Depression in Rural Veterans With Parkinson's Disease
Brief Title: Behavioral Treatments for Anxiety and Depression in Veterans With Parkinson's Disease
Acronym: BehTA-D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jessica Calleo, Clinical Psychologist, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28002
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson Disease; Anxiety; Depression
Keywords: Parkinson Disease; Anxiety; Depression
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — A modified version of existing Cognitive Behavioral Treatment and Self-management manuals.

SUMMARY:
Behavioral Treatments for Anxiety and Depression (BehTA-D) is a research study for anxiety and depression in individuals with Parkinson's disease (PD). The research clinicians try to teach skills that may help participants cope with anxiety and depression in the context of Parkinson's disease. Research clinicians will also discuss ways improve management of Parkinson's symptoms. Other skills taught include how to relax, change thinking, add in meaningful pleasant activity.

DETAILED DESCRIPTION:
Components of evidence-based cognitive behavioral therapy (CBT) treatments from current manuals developed for depression and anxiety will be used to construct the 8-week treatment program. The flexibility of modular based treatment allows patients and counselors to personalize interventions and skills for managing anxiety and depressive symptoms. The first treatment session will be in-person. All following sessions will be provided by telephone. Caregivers will have the option of being involved in 2 ways throughout treatment - as a "coach" to facilitate use of new skills by their loved one with PD and as a recipient of stress- management support. The scope of caregiver involvement will vary across patients, based on their preference. Involved caregivers will be given the opportunity to participate in 1 telephone-based stress-management session and 1 follow-up call scheduled individually during the first 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of idiopathic Parkinson's disease
2. Have significant anxiety and/or depressive symptoms as indicated by a score of greater than 4 on the Geriatric Depression Scale -15 or greater than 5 on the Hospital Anxiety and Depression anxiety subscale

Exclusion Criteria:

Patients will be excluded if they have cognitive impairment as indicated by the Montreal Cognitive Assessment (MoCA < 23) or if they have a condition that threatens their safety or life including suicidal intent, current psychosis, bipolar, substance abuse or impulse control disorders within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale and Hamilton Anxiety Scale | Baseline, 3-months and 4-months
Hamilton Depression Scale and Geriatric Depression Scale - 15 | Baseline, 3-months, and 4-months

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire -8 | Baseline, 3-months and 4-months
Client Satisfaction Questionnaire | 3-months and 4-months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica S Calleo, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey Veteran Affairs Medical Center, Houston, Texas, United States